CLINICAL TRIAL: NCT01163708
Title: Phase IV Study - Prophecy Guide Outcomes in Total Knee Replacement Surgery
Brief Title: Prophecy Guide Outcomes in Total Knee Replacement Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Global Orthopaedic Technology (Industry)
Collaborators: LSS Surgical Pty Ltd (Unknown)
Responsible Party: Dr Hugh English - Principal Investigator, Brisbane Orthopaedic Specialist Services
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Pro-Nav-10
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Osteoarthritis of the Knee; Total Knee Replacement
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Surgical Navigation Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigation alone (Active Comparator): Navigation system alone vs Prophecy technique with Navigation system validation
  Interventions: Device: Navigation System
- Prophecy and Navigation validation (Experimental)
  Interventions: Device: Prophecy Technique

INTERVENTIONS:
Device: Prophecy Technique — Navigation computerised system is used intraoperatively to correct implant the Advance knee implant. Prophecy is a pre-alignment technique where a pre-op MRI or CT scan is used to manufacture personalised cutting blocks to assist the surgeon in correct implanting the Advance knee implant intraoperatively
  Other Names: Prophecy Preoperative alignment
  Arms: Prophecy and Navigation validation
Device: Navigation System
  Arms: Navigation alone

SUMMARY:
This project aims to assess two different techniques used to position the knee replacement implant during surgery. The patients will be randomised to receive either the following:

1. The established Navigation System (gold standard)
2. The new Prophecy Technique (validated by the Navigation System)

The study hypothesis is there will be no difference between the gold standard Navigation system and the Prophecy technique in relation to the placement of the knee implant.

DETAILED DESCRIPTION:
Knee joint pain is often the cause of reduced joint and limb function. Total knee joint replacement is a procedure which aims to relieve pain and help to improve mobility. There has been continued development and improvement in knee implant design and the instruments required during surgery to assist with the accurate placement of the implant. These developments have reduced surgery time and assisted in the accurate positioning of the knee implant, which leads to better long term outcomes.

Navigation system is a computerised system currently used intraoperatively to position the Advance knee implant. The Prophecy technique is a pre-operative alignment technique. Patient undergo a MRI or CT scan which is used to manufacture personalised cutting blocks which are then used intraoperatively to position the knee implant.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring a total Knee Arthroplasty as determined jointly by the surgeon and the patient.
2. Over 65 years of age at time of surgery.
3. Patients with the Varus or Valgus Osteoarthritis
4. Patients who understand the conditions of the study and are willing to participate for the length of the prescribed term of follow-up.
5. Patients who are capable of, and have given, informed consent to their participation in the study.
6. The individual does not have an active infection within the affected joint.
7. The individual has not had a previous total knee replacement or knee fusion of the affected knee joint.
8. The individual is skeletally mature.
9. The individual is not pregnant.
10. The individual is not a prisoner.
11. The individual has no plans to relocate to another geographic area before the completion of the study.

Exclusion Criteria:

1. Previous surgery requiring implanting a device.
2. Knee deformity is >30° anatomic varus (as measured on an AP radiograph taken with the patient standing)
3. Knee deformity is >30° anatomic valgus (as measured on an AP radiograph taken with the patient standing) >20° knee flexion contracture (as measured by investigator examination)
4. Those patients requiring bone grafting or any other procedure that would extend the operative time beyond that of just replacing the knee should be excluded.
5. The individual is classified as morbidly obese (>40 BMI).
6. The individual is physically or mentally compromised (i.e., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, presence of alcohol or substance abuse), and is unwilling or unable to comply with postoperative scheduled clinical and radiographic evaluation and rehabilitation.
7. The individual has a neuromuscular or neuro-sensory deficiency which limits the ability to evaluate the safety and effectiveness of the device.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2010-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Prophecy Guide Outcomes in Total Knee Replacement Surgery | 5 years
  The primary objective of this study is to investigate the Prophecy technique and compare its outcomes to the established navigation (Gold standard) technique

SECONDARY OUTCOMES:
Prophecy Guide Outcomes in Total Knee Replacement Surgery | 5 years
  The secondary objectives are to evaluate the:
  1. Post-Operative Knee Alignment
  2. Implant sizing
  3. Implant position
  4. Tourniquet time
  5. Anaesthesia time
  6. Duration of surgery
  7. Validation of Prophecy MRI protocol
  8. Validation of bone resection

CONTACTS AND LOCATIONS:
Overall Officials: Hugh English, Principal Investigator — Brisbane Orthopaedic Specialist Services
Locations (2):
- Australia (2):
  - Holy Spirit Northside Private Hospital, Chermside, Queensland
  - Prince Charles Hospital, Chermside, Queensland